CLINICAL TRIAL: NCT01134913
Title: Multi-Markers In the Diagnosis of Acute Coronary Syndrome - Sample Procurement Cohort 3
Brief Title: Multi-Markers In the Diagnosis of Acute Coronary Syndrome
Acronym: Midas 3
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Sponsor
Other Study IDs: BSTE-0101-1
Record Dates: First submitted 2010-05-29; First posted 2010-06-02 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS; Acute Coronary Syndrome; Emergency Department
MeSH Terms: conditions — Acute Coronary Syndrome; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA Plasma Specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective clinical study designed to procure blood samples from patients who present to the Emergency Department with suspected ACS (Acute Coronary Syndrome).

Subjects enrolled in this study will sign and informed consent and have 4 blood samples drawn at different time points during their emergency department visit. In addition, data will be collected about the patient's health history, hospital procedures, and final diagnosis. The enrolling center will also contact the patients at 30-days, 3 months and 6 months to inquire about their condition and survival.

Blood samples collected in this study will be sent to the sponsor organization for long-term storage and analysis in the future for novel blood markers as they become available. No genetic testing will be conducted on these samples.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational, and sample procurement study of adult subjects presenting to an Emergency Department (ED) in whom ACS is in the differential diagnosis. Subjects must present to one of the participating EDs within 6 hours or less from the time of symptom onset, and must have experienced at least 5 minutes of chest discomfort.

Those ED patients with possible ACS who meet the inclusion/exclusion criteria will be approached for study enrollment by trained research personnel.

The patient's diagnostic work-up and treatment will continue per the standards of the treating institution. As indicated by their clinical presentation, it is anticipated that all patients in this study will have an electrocardiogram (ECG) upon admission to the ED and if the patient is found not to have an ST-elevation myocardial infarction (STEMI), objective cardiac testing will be conducted for evidence of MI. The Principal Investigator at each site will evaluate the results of the objective cardiac tests combined with biomarker evidence of myocardial necrosis to determine whether or not a patient enrolled at their site has a final diagnosis of ACS.

Cardiac events and procedure, such as angioplasty-stenting and coronary artery bypass surgery (CABG), will be recorded during the index ED visit, hospitalization and post-hospital follow-up period. Subjects will have a 30-day, 3 month and 6 month follow-up contact by phone or medical chart review to collect this information on cardiac events, procedures and survival.

Blood samples collected at several time points during the index ED visit will be used for future testing of novel blood markers as they become available.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older at time of enrollment.
2. Patient presenting to the ED within 6 hours from the onset of symptoms consistent with ACS.
3. Subject presented with at least one symptom outlined below:

   1. Chest discomfort of at least 5 minutes duration from time of symptom onset. Episodic or stuttering chest discomfort is acceptable if last episode preceding the ED presentation is within 6 hours of symptom onset.
   2. Chest discomfort of shorter duration due to pharmacologic intervention.
   3. Ischemic Equivalent, Chest Pain Syndrome, Anginal Equivalent, or Ischemic ECG Abnormalities.
4. Physician plans to perform objective cardiac testing as defined by the protocol in Section 3.2.

Exclusion Criteria:

1. Patient (or Legal Representative) unable or unwilling to provide informed consent.
2. Patient (or Legal Representative) refusal of telephone follow-up or medical record review at 30 days, 90 days and 180 days post-ED presentation.
3. Patient (or Legal Representative) refusal for multiple blood sample collections over the study period.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the ED within 6 hours with symptoms consistent with ACS.
Sampling Method: Non-Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Hospital, Boston, Massachusetts
  - New York Methodist Hospital, Brooklyn, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philidelphia, Pennsylvania

REFERENCES:
- [Derived] Smith SW, Diercks DB, Nagurney JT, Hollander JE, Miller CD, Schrock JW, Singer AJ, Apple FS, McCullough PA, Ruff CT, Sesma A Jr, Peacock WF. Central versus local adjudication of myocardial infarction in a cardiac biomarker trial. Am Heart J. 2013 Mar;165(3):273-279.e1. doi: 10.1016/j.ahj.2012.12.012. Epub 2013 Jan 26. PMID 23453092
- [Derived] Peacock WF, Nagurney J, Birkhahn R, Singer A, Shapiro N, Hollander J, Glynn T, Nowak R, Safdar B, Miller C, Peberdy M, Counselman F, Chandra A, Kosowsky J, Neuenschwander J, Schrock J, Plantholt S, Lewandrowski E, Wong V, Kupfer K, Diercks D. Myeloperoxidase in the diagnosis of acute coronary syndromes: the importance of spectrum. Am Heart J. 2011 Nov;162(5):893-9. doi: 10.1016/j.ahj.2011.08.017. PMID 22093206